CLINICAL TRIAL: NCT05363436
Title: Successful Implementation of an Opioid Reduction Toolkit in Pancreatectomy Patients Significantly Decreases Number of Opioids Prescribed and Consumed
Brief Title: Opioid Reduction Toolkit Reduces Opioids Prescribed and Consumed
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment Reorganzing
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19D.688Panc
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Opioid Abuse; Opioid Misuse; Pain
MeSH Terms: conditions — Opioid-Related Disorders; Pain | interventions — Oxycodone

STUDY DESIGN:
Intervention Model Description: Control group, measurement, intervention group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Normal Standard Practices of Prescribing
- Intervention (Experimental): Providers prescribed a base of 15 narcotic pills
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — Providers had to prescribe 15 oxycodone pills to each patient discharge
  Arms: Intervention

SUMMARY:
Investigators studied a baseline population of patients receiving pancreatectomies at their institution and determined how many opioid pills each patient was prescribed and how many they took. Based on this data they created a toolkit to provide to prescribers to give patients a modified number of pills. The amount prescribed and consumed was measured after intervention.

DETAILED DESCRIPTION:
A single academic surgical department reviewed opioid treatment patterns for patients undergoing common procedures, including open pancreatectomy, and an opioid reduction toolkit using the data collected was created. Providers were educated on the use of the toolkit and it was implemented as a standard of practice. Data were collected on pancreatectomy patients via telephone interview (performed at 2 weeks post-op) and by reviewing the state prescription drug monitoring program. Outcome variables included morphine milliequivalents (MME) of pills prescribed, MME of pills consumed, number of patients aware of proper unused pill disposal, number of patients requesting refills, and pain scores. Categorical and continuous outcomes were compared within and between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Being scheduled for an outpatient elective pancreatectomy

Exclusion Criteria:

* Urgent/emergent status
* Concomitant procedure being performed at time of pancreatectomy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of opioid pills reported being taken by the patient | 14 days
  Patients will be interviewed fourteen days after procedure and asked how many opioid pills they have taken since being discharged form the hospitals
Number of opioid pills being prescribed | 14 days
  Discharge paperwork and prescription information will be searched to determine the number of opioid pills were provided to the patient at discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No